CLINICAL TRIAL: NCT05364294
Title: Molecular Diagnosis of Systemic Autoinflammatory Diseases
Acronym: SAIDiag
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-97
Record Dates: First submitted 2022-04-08; First posted 2022-05-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Inflammatory Disease; Genetic Disease; Somatic Mutation; Molecular Sequence Variation; Molecular Pathway Deregulation
Keywords: Biomarkers
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Collectionof blood samples in a cohort of SAIDs patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Systemic autoinflammatory diseases (SAIDs) are a set of rare clinically and genetically heterogeneous conditions. The project proposes to identify novel genes and specific signatures in subgroups of patients with SAIDs.

DETAILED DESCRIPTION:
SAIDs are characterized by long dormant periods with no or only minor clinical symptoms interrupted by febrile crises accompanied by serous and synovial membrane inflammation that spontaneously resolves. Over the last decades, more than 50 genes encoding key components of the innate immune system have been identified to be involved in the pathophysiology of SAIDs, with both germline and somatic mosaic variations. When disease-causing variations are identified, specific biotherapies are proposed depending on the involved gene and pathway. However, despite these scientific advances, most SAIDs (70%) are of unknown etiology, the diagnosis is made with significant delay, and no targeted therapy can be suggested. This project aims to generate specific understanding and develop strategies for SAID patients with unknown etiology. The investigators aim to advance our understanding of SAIDs pathophysiology, find the disease-causing gene variations and identify the involved cellular pathways that should accelerate correct diagnosis and personalize treatment.

ELIGIBILITY:
Inclusion Criteria:

* A patient presenting with a clinical and biological aseptic inflammatory syndrome associating one or more of the following signs: spontaneously resolving fever, abdominal (pain, diarrhea), locomotor (arthralgia, myalgia), thoracic (pain, pericarditis), cutaneous, sensory (uveitis, deafness), or renal (amyloidosis) involvement.

Exclusion Criteria:

* Adult subject to legal protection measures (guardianship, curatorship, safeguard of justice).

Ages: 1 Week to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants in this research will be recruited during a follow-up consultation for their condition.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2032-05-31 (Estimated); Study Completion 2033-05-02 (Estimated)

PRIMARY OUTCOMES:
To identify SAIDs disease-causing mutations and genes and to explore specific biological signatures. | Anytime in the period of 10 years
  Molecular studies will be performed through the use of a SAID next generation sequencing (NGS) gene panel, followed by whole exome/genome sequencing (WES/WGS) in patients with no obvious genetic abnormality identified by the gene panel. When possible trio studies (the patient and his parents) will be performed in order to facilitate the interpretation of the molecular variants. Transcriptomics and cytokines profiles will be performed on whole blood cells to identify weakly expressed genes/proteins and by single cell experiments in order to assess cell-specific expression. These data will permit to better shape functional studies and to explore specific biological signatures.
To identify novel and better assess the disease pathways | Anytime in the period of 10 years
  Functional studies will be performed to evaluate the pathogenicity of the identified molecular variants, to assess the involvement of new candidate genes in SAIDs, to characterize the molecular networks to which the corresponding proteins belong and to open up new therapeutic avenues.

SECONDARY OUTCOMES:
To propose personalized treatment options | Anytime in the period of 10 years
  Depending on the disease gene identified and on the involved signalling pathway, specific biotherapies could be proposed to SAID patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Trousseau Hospital, Paris, France